CLINICAL TRIAL: NCT05175521
Title: Double Blind Randomized Control Trial of Inhaled Isopropyl Alcohol Vapors Versus Inhaled Eucalyptus Scent for the Treatment of Nausea Associated With Acute Migraine
Brief Title: Inhaled IAV vs Inhaled Eucalyptus for the Treatment of Nausea With Acute Migraine
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HonorHealth Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1718502
Record Dates: First submitted 2021-08-19; First posted 2022-01-03 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Migraine
Keywords: Nausea; Isopropyl alcohol; Eucalyptus; Aromatherapy; Vapors
MeSH Terms: conditions — Migraine Disorders; Nausea | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eucalyptus Oil Scent (Placebo Comparator): Eucalyptus oil diluted in mineral oil 1:20
  Interventions: Other: Eucalyptus Oil Scent
- Isopropyl Alcohol Vapors (Active Comparator): Isopropyl Alcohol 70%
  Interventions: Other: Isopropyl Alcohol Vapors

INTERVENTIONS:
Other: Eucalyptus Oil Scent — Eucalyptus oil in mineral (1:20) will be inhaled at least 30 minutes after onset of nausea associated with a migraine attack
  Arms: Eucalyptus Oil Scent
Other: Isopropyl Alcohol Vapors — Isopropyl Alcohol 70% will be inhaled at least 30 minutes after onset of nausea associated with a migraine attack
  Arms: Isopropyl Alcohol Vapors

SUMMARY:
The goal of this study is to compare the efficacy and adverse events of inhaled isopropyl alcohol vapor (IAV) versus placebo (inhaled eucalyptus scent (IES) (1:20 dilution in mineral oil) for treating nausea associated with acute migraine attacks.

DETAILED DESCRIPTION:
The main goal of this study is to examine the efficacy of (nausea reduction and time to use of other anti-nausea medications) and side effects of inhaled isopropyl alcohol vapor (IAV) for treating nausea among migraine patients using a double blind randomized control methodology. IAV is being compared inhaled eucalyptus scent (IES) (1:20 dilution in mineral oil) which has not shown benefit for treating nausea or migraine and is therefore considered placebo in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 to 65 years old with nausea associated migraines at least twice per month

Exclusion Criteria:

* Patients <18 or >65 years old
* Patients without a diagnosis of acute migraine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change of Severity of Nausea on Nausea Scale | ½ hour or to the end of treatment
  Change in Nausea, modified visual analog score from 0-10 with 10 severe nausea with vomiting, 5 moderate nausea, 1 mild nausea and 0 no nausea.

SECONDARY OUTCOMES:
Side effects associated with interventional substance | ½ hour, but likely less than 2 hours
  Patient written report
Use of anti-nausea medication/Time to use of anti-nausea medication | ½ hour or to the end of treatment
  Did using IAV vs eucalyptus oil change the time until use of oral anti-emetic?
Time to Clinically Relevant Nausea Change | ½ hour or to the end of treatment
  Did IAV vs eucalyptus oil reduce the amount of time the patient experienced nausea with their migraine?

CONTACTS AND LOCATIONS:
Overall Officials: Jill Rau, MD, PhD, Principal Investigator — HonorHealth Research Institute
Locations (1):
- HonorHealth Bob Bové Neuroscience Institute, Scottsdale, Arizona, United States